CLINICAL TRIAL: NCT05669937
Title: Turkish Validity and Reliability of the Baby Preparation and Worry Scale
Brief Title: Validity and Reliability of the Baby Preparation and Worry Scale
Status: Completed | Type: Observational
Sponsor: Mevlüde Alpaslan Arar (Other)
Responsible Party: Sponsor-Investigator, Mevlüde Alpaslan Arar, nurse, Ordu University
Organization: Ordu University (Other)
Other Study IDs: eylül2
Record Dates: First submitted 2022-11-30; First posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Mothers
Keywords: Infant Preparation; Worry; Mother health; Assessment Tool; Validity and Reliability,

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Reliable and valid measurement tools are needed to capture key components of prenatal distress, including anxiety and anxiety states that may put women and children at increased risk in the postpartum period.

Aim: The aim of this study is to determine the validity and reliability of the Baby Preparation and Worry Scale (Baby-PAWS), by adapting it to Turkish culture.

.

ELIGIBILITY:
Inclusion Criteria:

- Women who were married, older than 18 years, at least primary school graduates, in the third trimester of pregnancy and who accepted participation in the study were included.

Exclusion Criteria:

- Pregnant women with chronic disease and psychiatric disease history were not included in the research.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: The population for this methodological study comprised pregnant women in the third trimester reached online through pregnancy platforms (Instagram, Facebook, pregnancy class WhatsApp groups, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
"Baby Preparation and Worry Scale (Baby-PAWS)" developed by Erickson et al. to Turkish culture and perform validity and reliability studies to contribute a new scale tool specific to this field to the literature | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Samsun, Turkey (Türkiye)